CLINICAL TRIAL: NCT06152263
Title: Color Information From Linked Color Imaging is Associated With Mucosal Microvascular Density in Chronic Atrophic Gastritis and Early Gastric Cancer
Brief Title: LCI in Chronic Atrophic Gastritis and Early Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: LCI in CAG and EGC
Record Dates: First submitted 2023-10-29; First posted 2023-11-30 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: CAG - Chronic Atrophic Gastritis; EGC - Early Gastric Cancer
Keywords: color information; linked color imaging; mucosal microvascular density; chronic atrophic gastritis; early gastric cancer
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endoscopic biopsy or resection will be performed, and the mucosal microvascular density will be histopathologically analyzed using the specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrophic or Cancerous: In each image, the color values of atrophic or cancerous will be quantified using the International Commission on Illumination 1976 (L∗, a∗, b∗) color space. Histological microvascular density in biopsy or resected specimens will be evaluated using CD31 immunostaining. Color differences at the atrophic border and cancerous border, defined as Euclidean distances of color values between the atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be calculated according to mucosal microvascular density.
  Interventions: Other: Compare color information and mucosal microvascular density
- Non-atrophic or Non-cancerous: In each image, the color values of non-atrophic or non-cancerous will be quantified using the International Commission on Illumination 1976 (L∗, a∗, b∗) color space. Histological microvascular density in biopsy or resected specimens will be evaluated using CD31 immunostaining. Color differences at the atrophic border and cancerous border, defined as Euclidean distances of color values between the atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be calculated according to mucosal microvascular density.

INTERVENTIONS:
Other: Compare color information and mucosal microvascular density — To investigate the association between the color and mucosal microvascular density of CAG and EGC using linked color imaging.
  Groups: Atrophic or Cancerous

SUMMARY:
Color change is a useful marker for the endoscopic identification of chronic atrophic gastritis (CAG) and gastric cancer (GC). Several histopathological studies have suggested a correlation between certain gastrointestinal lesions and intramucosal vascularity. The aim of this study is to investigate the association between the color and mucosal microvascular density of CAG and early GC using linked color imaging (LCI). In this study, Lesions diagnosed as CAG and early GC will be observed using LCI. In each image, the color values of atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be quantified using the International Commission on Illumination 1976 (L∗, a∗, b∗) color space. Histological microvascular density in biopsy or resected specimens will be evaluated using CD31 immunostaining. Color differences at the atrophic border and cancerous border, defined as Euclidean distances of color values between the atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be calculated according to mucosal microvascular density.

DETAILED DESCRIPTION:
In this study, 10 patients diagnosed with CAG or early GC by esophagogastroduodenoscopy at Fifth Medical Center of Chinese PLA General Hospital between September 2023 and December 2023 will be enrolled. The following equipment will be used for the study: LCI endoscope (EG-760Z, FUJIFILM Co., Tokyo, Japan), light sources (LASEREO LL-4450; Fujifilm Co.), and video processors (AdvanciaHD VP-4450HD; FUJIFILM Co.). During esophagogastroduodenography, the atrophic or cancerous border will be identified. Following identical compositions, images will be continuously captured via LCI. Endoscopic biopsy or resection will be performed, and the mucosal microvascular density will be histopathologically analyzed using the specimens. The color values of atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be quantified using the International Commission on Illumination 1976 (L∗, a∗, b∗) color space. Histological microvascular density in biopsy or resected specimens will be evaluated using CD31 immunostaining. Color differences at the atrophic border and cancerous border, defined as Euclidean distances of color values between the atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be calculated according to mucosal microvascular density.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic atrophic gastritis (CAG) and early gastric cancer (EGC). by esophagogastroduodenoscopy

Exclusion Criteria:

* Inappropriate LCI images as a result of bleeding, ulceration, or excessive mucosal congestion
* Patients with severe anemia or portal hypertension
* Patients diagnosed as having a mixture of the differentiated and undifferentiated types of gastric carcinoma, or having helicobacter pylori infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CAG or EGC by esophagogastroduodenoscopy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Color differences between the atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa | up to 4 weeks
  The color values of atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be quantified by using the International Commission on Illumination 1976 (L∗, a∗, b∗) color space. It is speculated that there is a significant difference in the color difference between atrophic and non-atrophic mucosa and between cancerous and non-cancerous mucosa.
Microvascular density differences between the atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa | up to 2 weeks
  Histological microvascular density of atrophic and non-atrophic mucosa, as well as cancerous and non-cancerous mucosa, will be evaluated by using CD31 immunostaining. It is speculated that there is a significant difference in the mucosal microvascular density between atrophic and non-atrophic mucosa and between cancerous and non-cancerous mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — The Fifth Medical Center of Chinese PLA General Hosptial
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No